CLINICAL TRIAL: NCT06489873
Title: The Role of Lutein, Zeaxanthin, and Fish Oil on Cognitive Function and Bone Health in Healthy Adults
Brief Title: Lutein, Zeaxathin, and Fish Oil Supplementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Allen Foundation Inc. (Other)
Responsible Party: Principal Investigator, Karen Beathard, Instructional Associate Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024-0035
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Performance; Age-Related Macular Degeneration; Bone Loss
Keywords: Lutein; Zeaxanthin; Fish Oil; Supplement; Macular Pigment; Macular Pigment Optical Density; Cognition; Age-related Macular Degeneration; Cognitive Performance
MeSH Terms: conditions — Macular Degeneration; Bone Diseases, Metabolic | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an LZF or placebo supplement group and asked to take the assigned supplement daily for six months.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A researcher not participating in the research randomized participants and packaged LZF and placebo supplements in the exact same bottle other than the participant number and delivered these to the PI for distribution. Only this person has the list of numbers associated with the supplements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LZF Supplement (Active Comparator): Participants will take one LZF supplement daily for six months.
  Interventions: Dietary Supplement: Active Comparator (Lutein, zeaxanthin, and fish oil supplement (LZF)
- Placebo (Placebo Comparator): Participants will take on placebo supplement daily for six months.
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Active Comparator (Lutein, zeaxanthin, and fish oil supplement (LZF) — Each participant will be assigned to t a LZF supplement daily for six months
  Arms: LZF Supplement
Dietary Supplement: Placebo Comparator — Each participant will be assigned to take a placebo supplement daily for six months
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn the impact of lutein, zeaxanthin, and fish oil (LZF) supplementation in healthy adults.

The main question it aims to answer is: Will supplementation with LZF improve macular pigment optical density (MPOD), cognitive performance and bone mass compared to controls after six months?

Subjects with an MPOD <.43 will significantly improve MPOD after 6-months of LZF supplementation.

Consuming a LZFO supplement for 6-months will improve visual cognitive performance. Consuming a LZFO supplement for 6-months will improve bone density.

Participants will be asked to take either a LZF supplement or placebo daily for 6 months.

DETAILED DESCRIPTION:
Macular degeneration, cognitive decline, and osteoporosis often occur with aging. Lutein, zeaxanthin, and fish oil (LZF) have been shown to have improvements in these areas. This 6-month double-blind randomized controlled trial will study the impact of LZF on cognitive performance, macular pigment optical density (MPOD), and bone health in healthy adults ages 18-45 with a MPOD <.43. We seek to create a precision nutrition model reducing macular degeneration, cognition, and bone health that includes non-invasive screening for high-risk carotenoid deficiencies (MPOD, dietary intake) and individual response to LZF supplementation.

Healthy adults ages 18-45 years with MPOD <.43 will be randomly assigned to take a LZF supplement with 7 mg lutein, 14 mg zeaxanthin, and 245 mg fish oil or a placebo daily for six months. They will have baseline and ending measures of fasting blood draw, MPOD, bone health using a DXA, and visual cognitive performance using Neurotracker software.

ELIGIBILITY:
Inclusion Criteria:

* <.43 MPOD, a self-reported best-corrected vision of 20/40 or better in each eye, a BMI range of 18.5-30, and meets the inclusion criteria on the preliminary participant questionnaire.

Exclusion Criteria:

* allergic to lutein, zeaxanthin, or fish oil, taking supplements with >6 mg lutein and/or >2 mg zeaxanthin for more than two months before study starts, MPOD between >.43, self-reported condition of vertigo, diabetic retinopathy, retinitis pigmentosa, optic neuropathy, retinal vascular occlusions, strabismus, autoimmune disorders related to visual health, currently pregnant or trying to become pregnant, history of concussion, vegan (due to gelatin in the placebo), and/or taking neuroactive medications, such as Ritalin, Adderall, antidepressants, etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Macular Pigment Optical Density (MPOD) | MPOD will be measured at baseline, 3 months after the start of the study, and at the final 6 month visit, which will be the completion of the study.
  The MPS II will be used to measure MPOD
Cognitive Performance | Cognitive performance will be measured at the three baseline appointments, the three appointments at 3 months, and the 3 appointments at 6 months after the start of the study, which will be the completion of the study
  Neurotracker 3-dimensional software will be used to measure cognitive performance. Each cognitive performance session will include 15 6-second tests that will establish a speed threshold.
Bone Density | Bone density will be measured at baseline and at the final 6 month visit, which will be the completion of the study.
  The Horizon™ DXA System will be used for rapid, dual-energy bone density measurements in a single-sweep.

SECONDARY OUTCOMES:
Lutein and Zeaxanthin Serum Levels | Serum lutein and zeaxanthin will be measured at baseline and at the final 6 month visit, which will be the completion of the study.
  Serum will be drawn and analyzed for lutein and zeaxanthin content

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Beathard, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Gilchrist Building, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No